CLINICAL TRIAL: NCT05808348
Title: Effect of COVID-19 On Pain, Fear of Falling, Fall Frequency, and Physical Activity Level in the Elderly
Brief Title: Effects of COVID-19 on the Elderly
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ozan Gür, PT, Research Assistant, Kırklareli University
Other Study IDs: E-35523585-302.99-75492
Record Dates: First submitted 2023-04-07; First posted 2023-04-11 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pain; Fear; Falling; Physical Activity; COVID-19; Aged
Keywords: COVID-19; Pain; Fear; Falling; Physical Activity; Aged
MeSH Terms: conditions — Pain; Motor Activity; COVID-19 | interventions — Weights and Measures; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Group: Demographic and clinical information, Numerical Pain Rating Scale, Falls Efficacy Scale International, Baecke Physical Activity Questionnaire
  Interventions: Other: Scales and questionnaires
- Healthy Group: Demographic and clinical information, Numerical Pain Rating Scale, Falls Efficacy Scale International, Baecke Physical Activity Questionnaire
  Interventions: Other: Scales and questionnaires

INTERVENTIONS:
Other: Scales and questionnaires — We will ask participants about their age, gender, height, weight, education level, medical history, number of falls in the last 1 year, status and length of COVID-19-related hospitalizations, and whether they have gotten the COVID-19 vaccine. The participants will be interviewed in person as part of the evaluation process.
  The Modified Baecke Physical Activity Questionnaire, the Fall Efficacy Scale-International, and the Numerical Pain Rating Scale will be used to assess the participants' levels of pain, fear of falling, and physical activity, respectively.

SUMMARY:
The goal of this observational study is to learn about in former COVID-19 patients. The main questions it aims to answer are:

* are there any association among pain, fear of falling, fall frequency, and physical activity level
* are there any difference between former COVID-19 elders and non-COVID-19 elderly population

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Being cooperative

Exclusion Criteria:

* Refusing to participate in the study
* Having significant vision and hearing problems
* Not completing the study questions

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: The study will be carried out with people aged 65 and over living in Kırklareli/Turkey. Individuals will be divided into 2 groups as the COVID-19 group and the control group, according to whether they have had COVID-19 infection in the last 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Fear of Falling | through study completion, an average of 6 months
  Falls Efficacy Scale - International (total score between 16-64) (higher values indicate higher fear of falling)

SECONDARY OUTCOMES:
Pain Regions and Pain Severity | through study completion, an average of 6 months
  Numerical Pain Rating Scale (total score between 0-10) (higher values indicate higher pain)
Fall Frequency | through study completion, an average of 6 months
  Fall Frequency in 1 year
Physical Activity Level | through study completion, an average of 6 months
  Baecke Physical Activity Questionnaire (total score between 3-15) (higher values indicate higher physical acitivity level)

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided